CLINICAL TRIAL: NCT01975077
Title: A Randomized, Open-label Phase Ib Trial of Fruquintinib "4mg Once Daily Continuous"Versus "5mg Once Daily 3wks on/1wk Off" in Patients With Metastatic Colorectal Carcinoma as 3rd Therapy
Brief Title: A Phase Ib Study of Fruquintinib in 3rd Line mCRC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: Fudan University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-013-00CH3
Record Dates: First submitted 2013-09-29; First posted 2013-11-04 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: patients with mCRC who failed 2nd therapy or more
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A- 4mg QD (Experimental): arm A- fruquintinib 4mg once daily, p.o.,continuous;given in 28-days cycles until disease progress, intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: fruquintinib
- B- 5mg once daily, 3wks on/1wk off (Experimental): arm B-fruquintinb 5mg once daily,p.o.,3 weeks on/1 week off, given in 28-day cycles until disease progress,intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: fruquintinib

INTERVENTIONS:
Drug: fruquintinib — Fruquintinib is a capsule in the form of 1mg and 5mg, orally, daily
  Other Names: HMPL-013

SUMMARY:
Fruquintinib is a novel oral small molecule compound discovered and developed by Hutchison MediPharma that selectively inhibits vascular endothelial growth factor receptors (VEGFR) 1, 2, and 3 and has demonstrated potent inhibitory effects on multiple human tumor xenografts.Based on first-in-human study, both 4mg QD and 5mg 3wks on/1wk off are safety and efficacy, this phase Ib study is to evaluable the safety, tolerability and efficacy of these 2 regimens with mCRC failed 2nd therapy or more and to determine the recommended dose and regimen in phase II/III study.

DETAILED DESCRIPTION:
This is a phase Ib, randomize, interventional, open-label, multicenter study to provide fruquintinib to subjects diagnosed with metastatic colorectal cancer who have failed after standard therapy and for whom no therapy alternatives exist.

The primary endpoint of this study will be safety.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 70 years of age , with ≥ 40Kg
* Histological or cytological confirmed colorectal cancer
* ECOG performance status of 0-1
* Standard regimen failed or no standard regimen available
* Adequate hepatic, renal, heart, and hematologic functions
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan)
* Signed and dated informed consent.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure

Exclusion Criteria:

* Pregnant or lactating women
* Any factors that influence the usage of oral administration
* Evidence of CNS metastasis
* Intercurrence with one of the following: non-controlled hypertension, coronary artery disease, arrhythmia and heart failure
* Abuse of alcohol or drugs
* Less than 4 weeks from the last clinical trial
* Previous treatment with VEGFR inhibition
* Disability of serious uncontrolled intercurrence infection
* Proteinuria ≥ 2+ (1.0g/24hr)
* Uncontrolled hemorrhage in GI
* Within 12 months before the first treatment occurs artery/venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack) etc.
* Within 6 months before the first treatment occurs acute myocardial infarction, acute coronary syndrome or CABG
* Bone fracture or wounds that was not cured for a long time
* Coagulation dysfunction, hemorrhagic tendency or receiving anticoagulant therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | from day 1 of first dosing to 30days after permanent discontinuation of HMPL-013
  The primary objective is evaluation of safety and tolerabilty with 2 regimens. The primary endpoint is the incidence of AEs, SAEs, Gr3/4 AEs and AEs led to dose interruption and dose discontinued

SECONDARY OUTCOMES:
objective response rate(ORR) | every 8 weeks until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months
  using RECIST version 1.1
pharmacokinetic profiles | Day 1-84 steady state
  At QD regimen, PK sampling will include a pre-dose and at the 1,2,4,8,24 hour time points on day 1 and day 21;a pre-dose and at the 2 hour time point on day 28,42,70,84.
  At 3wks on/1wk off regimen,PK sampling will include a pre-dose and at the 1,2,4,8,24 hour time points on day 1 and day 21; a pre-dose and at the 2 hour time point on day 42 and day 70; only pre-dose on day 28,56,84.
disease control rate (DCR) | every 8 weeks until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months
  using RECIST version 1.1
progression-free survival (PFS) | every 8 weeks until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months
  using RECIST version 1.1
overall survival (OS) | every 2 months since end of treatment
  from first dosing until death due to any cause, assessed up to 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Fudan University Cancer Center, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Xu RH, Li J, Bai Y, Xu J, Liu T, Shen L, Wang L, Pan H, Cao J, Zhang D, Fan S, Hua Y, Su W. Safety and efficacy of fruquintinib in patients with previously treated metastatic colorectal cancer: a phase Ib study and a randomized double-blind phase II study. J Hematol Oncol. 2017 Jan 19;10(1):22. doi: 10.1186/s13045-016-0384-9. PMID 28103904